CLINICAL TRIAL: NCT05728125
Title: An In Depth Study Evaluating The Experiences of Patients In Glioblastoma Clinical Trials
Brief Title: Pinpointing the Factors Affecting Clinical Trial Experiences of Glioblastoma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 82966461
Record Dates: First submitted 2023-02-04; First posted 2023-02-14 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Glioblastoma
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Historically, clinical study participation has been biased toward certain demographics. However, there is a shortage of studies that delve into the underlying factors that influence patient participation, both positively and negatively.

Several people will be invited to enroll in this study so that it may collect a variety of data about glioblastoma clinical trial experiences and identify barriers to participation as well as the causes of participants' failure or withdrawal.

The data collected from this study will be analyzed and used to improve the experiences of future glioblastoma patients who are recruited for medical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patient has self-identified as planning to enroll in a clinical trial
* Patient has been diagnosed with glioblastoma
* Patient is a minimum of 18 years or older

Exclusion Criteria:

* Patient does not understand, sign, and return consent form
* Inability to perform regular electronic reporting
* Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glioblastoma patients who are actively considering enrolling in an observational clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to participate in a glioblastoma clinical trial | 3 months
Rate of patients who remain in glioblastoma clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wirsching HG, Galanis E, Weller M. Glioblastoma. Handb Clin Neurol. 2016;134:381-97. doi: 10.1016/B978-0-12-802997-8.00023-2. PMID 26948367
- [Background] Omuro A, DeAngelis LM. Glioblastoma and other malignant gliomas: a clinical review. JAMA. 2013 Nov 6;310(17):1842-50. doi: 10.1001/jama.2013.280319. PMID 24193082
- [Background] Luo C, Song K, Wu S, Hameed NUF, Kudulaiti N, Xu H, Qin ZY, Wu JS. The prognosis of glioblastoma: a large, multifactorial study. Br J Neurosurg. 2021 Oct;35(5):555-561. doi: 10.1080/02688697.2021.1907306. Epub 2021 Jul 8. PMID 34236262

DOCUMENTS (1):
  • Informed Consent Form (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT05728125/ICF_000.pdf